CLINICAL TRIAL: NCT03522350
Title: Randomized Controlled Trial Comparing EmbryoScope Time-Lapse System With the New Model EmbryoScope+.
Brief Title: Randomized Trial Comparing EmbryoScope With EmbryoScope+.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device has been FDA approved.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1612017837
Record Dates: First submitted 2018-02-20; First posted 2018-05-11 (Actual); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Infertility
Keywords: Infertility; Embryo develpoment; IVF; ICSI; EmbryoScope
MeSH Terms: conditions — Infertility | interventions — Fetoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- EmbryoScope (Active Comparator): Standard of care embryo incubator.
  Interventions: Device: EmbryoScope
- EmbryoScope+ (Experimental): New experimental embryo incubator.
  Interventions: Device: EmbryoScope+

INTERVENTIONS:
Device: EmbryoScope — Standard of care arm
  Arms: EmbryoScope
Device: EmbryoScope+ — Experimental arm
  Arms: EmbryoScope+

SUMMARY:
The purpose of the study is to compare the current EmbryoScope Time-Lapse System being used in IVF which has become standard of care to the new model EmbryoScope to demonstrate that the EmbryoScope+ is as safe and reliable as the EmbryoScope.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-center study in otherwise healthy infertile female subjects undergoing in vitro fertilization (IVF). The subjects recruited for this study will be among those patients who have been diagnosed with infertility and are planning to undergo IVF at the center where this study is being performed. The subjects will have undergone the usual informed consent procedure at the center.

Subjects will undergo ovarian stimulation, oocyte retrieval, IVF, and Intra Cytoplasmic Sperm Injection (ICSI) procedure following the center's usual procedures. At the time of retrieval, participant's oocytes will be randomly assigned to both groups for comparison: Standard EmbryoScope Time-Lapse system versus EmbryoScope+. The best quality embryos are selected for embryo transfer and the pregnancy outcome is evaluated.

"Best grade" embryos will be transferred regardless of EmbryoScope use. The standard EmbryoScope as well as the EmbryoScope+ monitor system as assigned during the randomization process will be used to observe the embryo development and document timing of embryo cleavages and morphology dynamics. Subjects will not be provided with the time- lapse images.

Endpoints will be Day 3 and Day 5/6 embryo development, implantation and pregnancy rate. The study is approximately 2 months, the estimated time it takes a physician to perform one IVF-ART treatment cycle. If embryos are frozen, the patient may be in the study until the time they choose to thaw the embryos or up to 1 year if they become pregnant.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or younger (maternal)
* 65 years of age or younger (paternal)
* Fresh or frozen (including donor) sperm can be used
* Fresh oocytes only (including donor)
* Frozen embryos from this study can be included in the outcome portion of this study.
* Single or double Blastocyst transfer only

Exclusion Criteria:

* 3 or more previous failed cycles
* Sperm obtained by testicular biopsy
* Co-culture patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Maternal age- 40 years of age or younger Paternal age- 65 years of age or younger
Enrollment: 18 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikica Zaninovic, PhD, Principal Investigator — Center for Reproductive Medicine
Locations (1):
- Center for Reproductive Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing IVF were be recruited to participate in the study. Those agreeing to participate consented to have their embryos incubated in the new Embryoscope+ as opposed to the current one being used as standard of care.
Pre-assignment Details: 18 subjects will undergo IVF. Participant's oocytes at retrieval will be randomly assigned to both groups for comparison: Standard EmbryoScope system versus EmbryoScope+. The best quality embryos are selected for embryo transfer and the pregnancy outcome is evaluated. "Best grade" embryos will be transferred regardless of EmbryoScope use.
Units Other Than Participants: Oocytes
Groups:
- Embryoscope +: Embryoscope +
- Embryoscope: Embryoscope
Period: Overall Study
Arm/Group | Embryoscope + | Embryoscope
Started | 18; 115 Oocytes | 18; 116 Oocytes
Completed | 18; 115 Oocytes | 18; 116 Oocytes
Not Completed | 0; 0 Oocytes | 0; 0 Oocytes

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This includes all participants - oocytes were randomized to standard of care embryo incubator and experimental Embryoscope +
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 33.6 [26 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Day 3 Embryos
Description: Comparing number of embryos that fertilized normally and had development at Day 3 based on embryo grade between oocytes assigned to Standard EmbryoScope versus oocytes assigned to EmbryoScope+
Time Frame: Day 3 post retrieval
Population: Number of day 3 embryos compared in both groups
Measure: Count of Units; unit: embryos
Units Other Than Participants: embryos
Arm/Group | Embryoscope + | Embryoscope
Number analyzed (Participants) | 18 | 18
Number analyzed (embryos) | 115 | 116
embryos | 42 | 42

2. Primary Outcome: Number of Day 5 Embryos
Description: Comparing the number pf embryos that developed at Day 5 based on embryo grade between oocytes assigned to Standard EmbryoScope versus oocytes assigned to EmbryoScope+
Time Frame: Day 5 post retrieval
Measure: Count of Units; unit: embryos
Units Other Than Participants: embryos
Arm/Group | Embryoscope + | Embryoscope
Number analyzed (Participants) | 18 | 18
Number analyzed (embryos) | 115 | 116
embryos | 43 | 51

3. Secondary Outcome: Implantation Rate
Description: Presence of a gestational sac
Time Frame: 5-6 weeks post retrieval
Measure: Count of Participants; unit: Participants
Arm/Group | Embryoscope + | Embryoscope
Number analyzed (Participants) | 18 | 18
Participants | 3 | 9

4. Secondary Outcome: Pregnancy Rate
Description: Positive Bhcg
Time Frame: 2 weeks post retrieval
Measure: Count of Participants; unit: Participants
Arm/Group | Embryoscope + | Embryoscope
Number analyzed (Participants) | 18 | 18
Participants | 4 | 9

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- All Participants Enrolled: All participants enrolled and randomized to Embryoscope and Embryoscope+
Arm/Group | All Participants Enrolled
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03522350/Prot_SAP_000.pdf